CLINICAL TRIAL: NCT01750359
Title: The Efficacy and Safety of Adjunctive Curcumin for Treatment of Depression: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety Curcumin in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vladimir Lerner (Other Government)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Sponsor-Investigator, Vladimir Lerner, A/Professor, Head of department, Beersheva Mental Health Center
Organization: Beersheva Mental Health Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LBM-2010; IsraelMHC (Other: Tirat Carmel &Be'er Sheva MHC)
Record Dates: First submitted 2012-07-25; First posted 2012-12-17 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2012-12

CONDITIONS: Major Depression
Keywords: antioxidants; curcumin; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcumin (Active Comparator)
  Interventions: Drug: curcumin
- placebo (Placebo Comparator)
  Interventions: Drug: curcumin

INTERVENTIONS:
Drug: curcumin — 500 mg/day for 6 week

SUMMARY:
Antidepressants generally do not lead to an immediate relief of symptoms. Most people will not see a significant improvement for at least 4 weeks. Studies have generally shown that the full benefits of antidepressant therapy may take as long as 8 to 12 weeks. However, this timeline is variable among individuals.Curcumin is one of the main curcuminoids isolated from this perennial herb. It possesses a variety of pharmacological activities, including anti-inflammatory, antiproliferative, antioxidant, and neuroprotective effects. Curcumin has been found to possess antidepressant action in various animal models of depression. Chronic administration of curcumin has been reported to exert antidepressant-like action in olfactory bulbectomy model of depression in rats. Although the mechanism of the antidepressant effect of curcumin is not fully understood, it is hypothesized that it acts through inhibiting the monoamine oxidase enzyme and modulating the release of serotonin and dopamine.In randomized, double-blind, placebo-controlled study 40 patients will be randomized to receive either 500 mg/day of curcumin or placebo together with antidepressants for 6 weeks.

ELIGIBILITY:
Inclusion criteria:

Males and females in age 20-60 years

Major depressive episode according to DSM-IV

Clinical Global Impression Severity Scale scores more than 4

Hamilton Depression Rating Scale scores more than 21

Montgomery and Asberg Depression Rating Scale scores more than 22

Ability and willingness to sign informed consent

Exclusion Criteria:

Evidence of organic brain damage

Mental retardation

Alcohol or drug abuse

An unstable medical condition

Any significant medical or neurological illness

Patients with a known hypersensitivity to curcumin or other components of the product

Pregnant women or women who intend to become pregnant

Receiving any antidepressant and mood-stabilizers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Change in the scores from baseline at six weeks
Montgomery-Asberg Depression Rating Scale | Change in the scores from baseline at six weeks

SECONDARY OUTCOMES:
Clinical Global Impression | Change in the scores from baseline at six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bergman, MD, Principal Investigator — Tirat Carmel; Vladimir Lerner, MD, PhD, Study Director — Beersheva Mental Health Center
Locations (1):
- Tirat Carmel Mental Health Center, Tirat Carmel, Israel